CLINICAL TRIAL: NCT06892028
Title: A Randomized Controlled Trial of Electroencephalogram (EEG) Personalized Transcranial Magnetic Stimulation (eTMS) for Post-Traumatic Stress Disorder
Brief Title: EEG-based Personalized Transcranial Magnetic Stimulation (eTMS) to Treat Post-Traumatic Stress Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: eTMS-PTSD-001-Stage 2; 2021 RFP # SRC2472 DMH009 (Other Grant/Funding Number: State of Ohio)
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Stress Disorder, Post Traumatic
Keywords: PTSD; Veterans; First Responders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active eTMS treatment (Active Comparator): 15 treatment days of EEG-based personalized TMS over a maximum of 28 days. Two sessions per treatment day. Each session consists of TMS treatment at 80% Motor Threshold, pulse frequency between 8-13 Hz. TMS delivery of 5 second pulse train, with an inter-train interval of 20 seconds. Session duration is 15 minutes. A rest period of at least 30 minutes is required between the 2 sessions in a treatment day.
  Interventions: Device: EEG-based personalized TMS
- Sham eTMS Treatment (Sham Comparator): 15 treatment days of sham EEG-based personalized TMS over a maximum of 28 days. Two sessions per treatment day. Each session consists of sham TMS treatment. TMS delivery of 5 second pulse train, with an inter-train interval of 20 seconds. Session duration is 15 minutes. A rest period of at least 30 minutes is required between the 2 sessions in a treatment day.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: EEG-based personalized TMS — Transcranial Magnetic Stimulation (TMS), in which treatment is personalized based on the participant's Electroencephalogram (EEG)
  Arms: Active eTMS treatment
Device: Sham Comparator — Sham Transcranial Magnetic Stimulation (TMS), in which treatment is personalized based on the participant's Electroencephalogram (EEG). No stimulation is provided.
  Arms: Sham eTMS Treatment

SUMMARY:
This is a randomized, sham controlled study of the Electroencephalogram (EEG) based Transcranial Magnetic Stimulation (eTMS) treatment for Post-Traumatic Stress Disorder (PTSD). The recruitment goal is 110 participants who are United States Military veterans or first responders (e.g., firefighters, police, paramedics, etc.). The Study includes an EEG recording in order to determine the optimal treatment parameters for the eTMS system, followed by 15 in-office visits that take place over 21-28 total days. Two eTMS treatment sessions are administered during each office visit.

DETAILED DESCRIPTION:
eTMS-PTSD-001 Stage 2 is a randomized, sham controlled study with a recruitment goal of 100 subjects, with 99 completers. The Study is intended to evaluate the safety and efficacy of eTMS in the target population. A maximum of 800 individuals will be screened in order to achieve the recruitment goal. The total number of days from the first participant enrolled to the last enrolled participant treated will be approximately 10 months.

Participants will be either Veterans or First Responders (e.g., emergency medical service provider, firefighter, or any other emergency response personnel), between 22-65 years of age. Participants may be male or female of any racial/ethnic background who meet the eligibility criteria. Participants will be recruited from the general public, and from veterans and first responder organizations.

The primary outcome for the Study will be reduction in PTSD symptoms as calculated by the PTSD Checklist for DSM-5 (PCL-5) assessment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to consent to participate in the study via signed Informed Consent
* Age 22 - 65 years
* Diagnosis of PTSD according to DSM-5 criteria via the Clinician-Administered PTSD Scale (CAPS).
* Onset of symptoms meeting the DSM-5 criteria for PTSD symptoms persisting for a minimum of 6 months prior to the Screening Visit
* Veterans Administration PCL-5 cut point score of 31 or above
* Positive identification as either a Veteran, or First Responder (e.g., emergency medical service provider, firefighter, or any other emergency response personnel)

Exclusion Criteria:

* Uncontrolled medical, psychological or neurological condition
* Pregnant, or female unwilling to use effective birth control during the course of the trial
* Metal objects in the head
* Past exposure to metal fragments, permanent piercings, and/or other possible metal sources in the head and neck
* Current participation in any interventional research protocol
* History of any type of Electroconvulsive Therapy (ECT) or repetitive Transcranial Magnetic Stimulation (rTMS)
* History of stroke or intracranial lesion or increased intracranial pressure
* History of epilepsy of seizure
* Family history of epilepsy or seizure in 1st degree relative
* An elevated risk of suicide or violence to others

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in PTSD Symptoms as Measured by Drop in Score on the PTSD Checklist for DSM-5 (PCL-5) | Baseline and Final Measure, between 21-28 Days
  The Post Traumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual of Mental Disorders, 5th Ed. (DSM-5), commonly referred to as PCL-5, is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. It is used to monitor symptom change during and after treatment. Each item is scored from 0 to 5 as the participant's estimate of the severity of the symptom (0 = Not at all, 1=A little bit, 2 = Moderately, 3 = Quite a bit, 4 = Extremely). The final score range is between 0-80. A lower score is considered better than a higher score.

SECONDARY OUTCOMES:
Number, Severity, Relatedness, Type, Subsequent Treatment/Intervention Required, and Resolution Status of Adverse Events (AEs) During the Study. | Baseline and Final Measure, between 21-28 Days
  Number - Number of adverse events reported. Note that each participant may have had more than one adverse event (AE).
  Severity - Number of adverse events that were mild, moderate, or severe. Relatedness - Number of adverse events that were not related, suspected, or definitely related to treatment.
  Type - Number of adverse events that were or were not Serious Adverse Events (SAEs).
  Subsequent treatment/intervention required - Number of adverse events that did or did not require subsequent treatment/intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Phillips, PhD, Principal Investigator — Wave Neuroscience, Inc.
Locations (2):
- United States (2):
  - Wright State University, Dayton, Ohio
  - D2 Human Performance Center, Pickerington, Ohio

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers

REFERENCES:
- [Background] Bae EH, Schrader LM, Machii K, Alonso-Alonso M, Riviello JJ Jr, Pascual-Leone A, Rotenberg A. Safety and tolerability of repetitive transcranial magnetic stimulation in patients with epilepsy: a review of the literature. Epilepsy Behav. 2007 Jun;10(4):521-8. doi: 10.1016/j.yebeh.2007.03.004. Epub 2007 May 9. PMID 17493877
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003388. doi: 10.1002/14651858.CD003388.pub3. PMID 17636720
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Caulfield KA. Is accelerated, high-dose theta burst stimulation a panacea for treatment-resistant depression? J Neurophysiol. 2020 Jan 1;123(1):1-3. doi: 10.1152/jn.00537.2019. Epub 2019 Sep 25. PMID 31553674
- [Background] Corlier J, Carpenter LL, Wilson AC, Tirrell E, Gobin AP, Kavanaugh B, Leuchter AF. The relationship between individual alpha peak frequency and clinical outcome with repetitive Transcranial Magnetic Stimulation (rTMS) treatment of Major Depressive Disorder (MDD). Brain Stimul. 2019 Nov-Dec;12(6):1572-1578. doi: 10.1016/j.brs.2019.07.018. Epub 2019 Jul 25. PMID 31378603
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Raman R, Benedek DM, Pelic CG, Grammer GG, Stokes KT, Schmidt M, Spiegel C, Dealmeida N, Beaver KL, Borckardt JJ, Sun X, Jain S, Stein MB. A two-site pilot randomized 3 day trial of high dose left prefrontal repetitive transcranial magnetic stimulation (rTMS) for suicidal inpatients. Brain Stimul. 2014 May-Jun;7(3):421-31. doi: 10.1016/j.brs.2014.03.006. Epub 2014 Mar 19. PMID 24731434
- [Background] George MS, Wassermann EM, Williams WA, Steppel J, Pascual-Leone A, Basser P, Hallett M, Post RM. Changes in mood and hormone levels after rapid-rate transcranial magnetic stimulation (rTMS) of the prefrontal cortex. J Neuropsychiatry Clin Neurosci. 1996 Spring;8(2):172-80. doi: 10.1176/jnp.8.2.172. PMID 9081553
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Hunter AM, Minzenberg MJ, Cook IA, Krantz DE, Levitt JG, Rotstein NM, Chawla SA, Leuchter AF. Concomitant medication use and clinical outcome of repetitive Transcranial Magnetic Stimulation (rTMS) treatment of Major Depressive Disorder. Brain Behav. 2019 May;9(5):e01275. doi: 10.1002/brb3.1275. Epub 2019 Apr 2. PMID 30941915
- [Background] Janicak PG, O'Reardon JP, Sampson SM, Husain MM, Lisanby SH, Rado JT, Heart KL, Demitrack MA. Transcranial magnetic stimulation in the treatment of major depressive disorder: a comprehensive summary of safety experience from acute exposure, extended exposure, and during reintroduction treatment. J Clin Psychiatry. 2008 Feb;69(2):222-32. doi: 10.4088/jcp.v69n0208. PMID 18232722
- [Background] Jin Y, Phillips B. A pilot study of the use of EEG-based synchronized Transcranial Magnetic Stimulation (sTMS) for treatment of Major Depression. BMC Psychiatry. 2014 Jan 18;14:13. doi: 10.1186/1471-244X-14-13. PMID 24438321
- [Background] Jin Y, Kemp AS, Huang Y, Thai TM, Liu Z, Xu W, He H, Potkin SG. Alpha EEG guided TMS in schizophrenia. Brain Stimul. 2012 Oct;5(4):560-8. doi: 10.1016/j.brs.2011.09.005. Epub 2011 Oct 6. PMID 22019083
- [Background] Leuchter AF, Cook IA, Jin Y, Phillips B. The relationship between brain oscillatory activity and therapeutic effectiveness of transcranial magnetic stimulation in the treatment of major depressive disorder. Front Hum Neurosci. 2013 Feb 26;7:37. doi: 10.3389/fnhum.2013.00037. eCollection 2013. PMID 23550274
- [Background] Loo CK, McFarquhar TF, Mitchell PB. A review of the safety of repetitive transcranial magnetic stimulation as a clinical treatment for depression. Int J Neuropsychopharmacol. 2008 Feb;11(1):131-47. doi: 10.1017/S1461145707007717. Epub 2007 Sep 20. PMID 17880752
- [Background] Loo C, Sachdev P, Elsayed H, McDarmont B, Mitchell P, Wilkinson M, Parker G, Gandevia S. Effects of a 2- to 4-week course of repetitive transcranial magnetic stimulation (rTMS) on neuropsychologic functioning, electroencephalogram, and auditory threshold in depressed patients. Biol Psychiatry. 2001 Apr 1;49(7):615-23. doi: 10.1016/s0006-3223(00)00996-3. PMID 11297719
- [Background] Machii K, Cohen D, Ramos-Estebanez C, Pascual-Leone A. Safety of rTMS to non-motor cortical areas in healthy participants and patients. Clin Neurophysiol. 2006 Feb;117(2):455-71. doi: 10.1016/j.clinph.2005.10.014. Epub 2006 Jan 4. PMID 16387549
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Background] Carpenter LL, Conelea C, Tyrka AR, Welch ES, Greenberg BD, Price LH, Niedzwiecki M, Yip AG, Barnes J, Philip NS. 5 Hz Repetitive transcranial magnetic stimulation for posttraumatic stress disorder comorbid with major depressive disorder. J Affect Disord. 2018 Aug 1;235:414-420. doi: 10.1016/j.jad.2018.04.009. Epub 2018 Apr 5. PMID 29677606
- [Background] Roelofs CL, Krepel N, Corlier J, Carpenter LL, Fitzgerald PB, Daskalakis ZJ, Tendolkar I, Wilson A, Downar J, Bailey NW, Blumberger DM, Vila-Rodriguez F, Leuchter AF, Arns M. Individual alpha frequency proximity associated with repetitive transcranial magnetic stimulation outcome: An independent replication study from the ICON-DB consortium. Clin Neurophysiol. 2021 Feb;132(2):643-649. doi: 10.1016/j.clinph.2020.10.017. Epub 2020 Nov 10. PMID 33243617
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Sakkas P, Mihalopoulou P, Mourtzouhou P, Psarros C, Masdrakis V, Politis A, Christodoulou GN. Induction of mania by rTMS: report of two cases. Eur Psychiatry. 2003 Jun;18(4):196-8. doi: 10.1016/s0924-9338(03)00048-8. PMID 12814856
- [Background] Wobrock T, Guse B, Cordes J, Wolwer W, Winterer G, Gaebel W, Langguth B, Landgrebe M, Eichhammer P, Frank E, Hajak G, Ohmann C, Verde PE, Rietschel M, Ahmed R, Honer WG, Malchow B, Schneider-Axmann T, Falkai P, Hasan A. Left prefrontal high-frequency repetitive transcranial magnetic stimulation for the treatment of schizophrenia with predominant negative symptoms: a sham-controlled, randomized multicenter trial. Biol Psychiatry. 2015 Jun 1;77(11):979-88. doi: 10.1016/j.biopsych.2014.10.009. Epub 2014 Oct 23. PMID 25582269
- [Background] Yesavage JA, Fairchild JK, Mi Z, Biswas K, Davis-Karim A, Phibbs CS, Forman SD, Thase M, Williams LM, Etkin A, O'Hara R, Georgette G, Beale T, Huang GD, Noda A, George MS; VA Cooperative Studies Program Study Team. Effect of Repetitive Transcranial Magnetic Stimulation on Treatment-Resistant Major Depression in US Veterans: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Sep 1;75(9):884-893. doi: 10.1001/jamapsychiatry.2018.1483. PMID 29955803
- [Background] Ziemann U. TMS and drugs. Clin Neurophysiol. 2004 Aug;115(8):1717-29. doi: 10.1016/j.clinph.2004.03.006. PMID 15261850
- [Background] Ziemann U, Reis J, Schwenkreis P, Rosanova M, Strafella A, Badawy R, Muller-Dahlhaus F. TMS and drugs revisited 2014. Clin Neurophysiol. 2015 Oct;126(10):1847-68. doi: 10.1016/j.clinph.2014.08.028. Epub 2014 Dec 4. PMID 25534482
- See also: Study Information Page — http://www.etmsfda.com